CLINICAL TRIAL: NCT04628000
Title: Baseline Vitamin D Deficiency and COVID-19 Disease Severity/Need for Escalation of Care
Brief Title: Baseline Vitamin D Deficiency and COVID-19 Disease Severity
Status: Completed | Type: Observational
Sponsor: Parkview Medical Center (Other)
Responsible Party: Principal Investigator, Doug Duffee, Research Committee Chair, Parkview Medical Center
Other Study IDs: PIRB78
Record Dates: First submitted 2020-11-11; First posted 2020-11-13 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Vitamin D Deficiency; Covid19
Keywords: prognosis
MeSH Terms: conditions — Vitamin D Deficiency; COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vitamin D deficiency and COVID19: Vitamin D deficiency and COVID19
  Interventions: Other: Vitamin D

INTERVENTIONS:
Other: Vitamin D — Clinical Correlation
  Other Names: Vitamin D deficiency

SUMMARY:
It is known that vitamin D has been found to decrease incidence of viral respiratory infections, as well as have effects on multiple cytokines involved in immunomodulation and the bradykinin/renin-angiotensin system.

Recently, data was released showing a correlation between baseline vitamin D deficiency status and increased risk of contracting COVID-19.

Separate analysis shows that many of the deleterious effects of COVID-19 may be due to the bradykinin/RAS system, and that vitamin D is one plausible treatment option to modulate these effects.

Studies are currently ongoing to determine if vitamin D supplementation of those hospitalized with COVID-19 has a beneficial effect on patient outcomes.

Healthcare resources have been strained during the pandemic in areas of heavy caseload. It is possible that those with concurrent vitamin D deficiency and COVID positivity have an increased need for escalation of care. A small study has been conducted in this area, but was limited by small number of subjects.

DETAILED DESCRIPTION:
Abstract: It is known that vitamin D has been found to decrease incidence of viral respiratory infections, as well as have effects on multiple cytokines involved in immunomodulation and the bradykinin/renin-angiotensin system. Recently, data was released showing a correlation between baseline vitamin D deficiency status and increased risk of contracting COVID-19. Separate analysis shows that many of the deleterious effects of COVID-19 may be due to the bradykinin/RAS system, and that vitamin D is one plausible treatment option to modulate these effects. Studies are currently ongoing to determine if vitamin D supplementation of those hospitalized with COVID-19 has a beneficial effect on patient outcomes.

Objective: To determine if those hospitalized with COVID-19 with baseline vitamin D deficiency, have worse outcomes during their stay than those who are not vitamin D deficient at baseline.

Design, Setting, and Participants: This is a retrospective cohort study at an urban academic medical center which included patients with a 25-hydroxycholecalciferol level measured within one year before being tested for COVID-19 and hospitalized from March 9th to September 7th, 2020.

Exposures: Vitamin D deficiency was defined by the last measurement of 25-hydroxycholecalciferol less than 20 ng/mL before COVID testing (within one year).

Main Outcomes and Measures: The primary outcomes investigated include length of stay, need for supplemental oxygen, ICU admission, need for invasive life support (mechanical ventilation, vasopressors, dialysis), and discharge status (discharged alive vs. death).

ELIGIBILITY:
Inclusion Criteria:

* Covid 19 +
* Vitamin D level

Exclusion Criteria:

* Age < 18
* no associated vitamin D level

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those hospitalized 3/9-9/7 2020 who were covid positive and had concomitant vit d level drawn
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
LOS duration in days | 3/9-9/7 2020
  Length of stay
Supp O2 flow volume in L/min | 3/9-9/7 2020
  Supplemental Oxygen need

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lucas, MD, Principal Investigator — Parkview Medical Center
Locations (1):
- Parkview Medical Center, Pueblo, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martineau AR, Jolliffe DA, Greenberg L, Aloia JF, Bergman P, Dubnov-Raz G, Esposito S, Ganmaa D, Ginde AA, Goodall EC, Grant CC, Janssens W, Jensen ME, Kerley CP, Laaksi I, Manaseki-Holland S, Mauger D, Murdoch DR, Neale R, Rees JR, Simpson S, Stelmach I, Trilok Kumar G, Urashima M, Camargo CA, Griffiths CJ, Hooper RL. Vitamin D supplementation to prevent acute respiratory infections: individual participant data meta-analysis. Health Technol Assess. 2019 Jan;23(2):1-44. doi: 10.3310/hta23020. PMID 30675873
- [Background] Grant WB, Lahore H, McDonnell SL, Baggerly CA, French CB, Aliano JL, Bhattoa HP. Evidence that Vitamin D Supplementation Could Reduce Risk of Influenza and COVID-19 Infections and Deaths. Nutrients. 2020 Apr 2;12(4):988. doi: 10.3390/nu12040988. PMID 32252338
- [Background] Garvin MR, Alvarez C, Miller JI, Prates ET, Walker AM, Amos BK, Mast AE, Justice A, Aronow B, Jacobson D. A mechanistic model and therapeutic interventions for COVID-19 involving a RAS-mediated bradykinin storm. Elife. 2020 Jul 7;9:e59177. doi: 10.7554/eLife.59177. PMID 32633718
- [Background] ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine (US). 2020 Apr 10 - . Identifier NCT04334005, Vitamin D on Prevention and Treatment of COVID 19 (COVITD-19) [cited 2020 Sept 9]; Available from: https://clinicaltrials.gov/ct2/show/NCT04334005